CLINICAL TRIAL: NCT04053530
Title: Evaluation of the Marginal Integrity of Recent Bulk Fill Flowable Composite vs Glass Ionomer for Carious Cervical Restorations: Randomized Controlled Clinical Trail
Brief Title: Evaluation of the Marginal Integrity of Recent Bulk Fill Flowable Composite vs Glass Ionomer for Carious Cervical Restorations: RCCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Reda Abd EL Rahman, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: oper 5215
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Dental Caries Class v

STUDY DESIGN:
Intervention Model Description: 3 parallel groups
Who Masked: Outcomes Assessor
Masking Description: Data analysts, statistician and outcome assessor (A.O.) will be blinded after assignment to interventions while the operator will not due to the difference in restorative material presentation and its application protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 3M™ Ketac™ Universal Aplicap™ (Experimental): 3M™ Ketac™ Universal Aplicap™ Glass Ionomer Restorative Clean the cavity preparation with water. Rinse thoroughly and dry. Extrude the mixed ketac universal out of the capsule directly into the prepared cavity with a capsule gun. Please ensure that no air bubbles are included.
  It is recommended that the finishing and polishing can be continued after approximately 4 minutes after the start of the mixing or earlier if heat is applied for faster setting. The finishing and polishing can be done immediately after final setting with Extra-Fine, Friction Grip diamonds under water-cooling.
  Interventions: Other: restorative materials
- Filtek™ Bulk Fill Flowable composite (Experimental): Filtek™ Bulk Fill Flowable Restorative is the 3M ESPE choice in the bulk fill flowable category.
  Selective etching 15-20 s for enamel. The adhesive system (BISCO universal all bond) will be applied following the manufacturer's instructions (apply 2 coats 20 s before curing). Bulk fill flowable composite will be light cured for 40 s using a visible light curing unit.
  Interventions: Other: restorative materials
- ketac N100 (Active Comparator): Ketac™ Nano Light Curing Glass Ionomer Restorative. Primer will be applied to both enamel and dentinal surfaces for 15 seconds. The prepared tooth surfaces will be wet with the primer for the full application time.
  Dispensing two clicks from the Clicker™ Dispenser will provide an adequate amount of material for most restorative filling applications.
  It will be placed with a syringe system then will be placed in 2mm increments or less, and light cured after each increment. An LED curing light will cure all shades with a 20 second light exposure.
  Finishing Ketac Nano restorative will be polished with conventional finishing and polishing instruments such as a diamond impregnated rubberized polishing system under water spray. A glaze such as Vitremer™ Finishing Gloss will be applied after polishing if desired.
  Interventions: Other: restorative materials

INTERVENTIONS:
Other: restorative materials — glass ionomer and bulk fill flowable composite

SUMMARY:
The study will be conducted to assess the marginal integrity of different types of restorations (ketac ™ N100 - ketac™ Universal and bulk fill flowable composite) in class v restoration using USPHS criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of at least one carious buccal cervical lesion.
2. The absence of tooth mobility.
3. Presence of contact with opposite teeth without any abnormal occlusion stress for the selected teeth.
4. Accessible isolation and observable and easily accessible gingival margins during tooth restoration.

Exclusion Criteria:

1. Patients with poor oral hygiene.
2. The presence of any para functional habit.
3. Abnormal occlusion.
4. Any regurgitation problem.
5. Subjects with compromised medical history.
6. Pulpitis, non-vital or endodontically treated teeth.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2019-08-04 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
is marginal integrity of restoration. | 12 months
  Primary outcome is marginal integrity of restoration. It will be assessed by USPHS; score will be recorded according to USPHS criteria (Nassar et al., 2014).
  1. MARGINAL INTEGRITY
  Alpha (A) Visual inspection and explorer The explorer does not catch when drawn across the surface of the restoration toward the tooth, or, if the explorer does not catch, there is no visible crevice along the periphery of the restoration.
  Bravo (B) Visual inspection and explorer The explorer catches and there is visible evidence of a crevice, which the explorer penetrates, indicating that the edge of the restoration does not adapt closely to the tooth structure. The dentin and/or the base is not exposed, and the restoration is not mobile.
  Charlie (C) Explorer The explorer penetrates crevice defect extended to the dentino-enamel junction.
  Delta (D) Mobile, fractured or missing restoration in a part or total

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo university, Cairo
  - Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: No